CLINICAL TRIAL: NCT01209715
Title: Effect of an Inhaled Glucocorticoid-long-acting Beta Adrenergic Agonist on Endothelial Function in COPD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the ubiquitous use of ICS in the treatment of COPD in 2012, it was hard to find the study population.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 114279
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: COPD
Keywords: airway blood flow,; COPD,; endothelial dysfunction; inhaled corticosteroids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matching Placebo (Placebo Comparator): Participants will be treated with placebo twice a day for 3 weeks.
  Interventions: Drug: Placebo; Drug: Fluticasone /salmeterol
- Fluticasone/salmeterol (Active Comparator): Participants will be assigned to inhaled fluticasone/salmeterol twice a day for 3 weeks.
  Interventions: Drug: Fluticasone /salmeterol

INTERVENTIONS:
Drug: Placebo — participants will be assigned to 3-weeks treatment of inhaled placebo twice a day
  Arms: Matching Placebo
Drug: Fluticasone /salmeterol — Participant will be assigned to a 3-weeks treatment with inhaled fluticasone/salmeterol or matching placebo
  Other Names: Advair 250/50

SUMMARY:
In the present study, the investigators wish to address the effect of a glucocorticoid/long-acting beta-agonist preparation on endothelial function in COPD patients who do not currently smoke (ex-smokers) by measuring endothelium-dependent (albuterol response) and endothelium-independent (NTG response) vasodilation in the bronchial artery, reflecting endothelium-dependent and endothelium-independent vasodilation (drug-induced increase in Qaw, ΔQaw). With this approach the investigators will test the hypothesis that in stable ICS-naïve COPD patients, endothelium-dependent vasodilation is restored with a glucocorticoid/long-acting beta-agonist preparation, presumably resulting from the glucocorticoid component.

DETAILED DESCRIPTION:
To test the premise and to characterize the time dependence of the responses, the investigators propose the following two aims:

1. To determine the effect of a medium dose glucocorticoid/long-acting beta-agonist preparation (250 μg fluticasone plus 50 μg salmeterol) administered for 3 weeks on inhaled albuterol and sub-lingual NTG induced vasodilation in the bronchial artery, as assessed by ΔQaw in stable glucocorticoid-naïve COPD patients, and to re-assess the responses after a 3 week glucocorticoid/long-acting beta-agonist washout period.
2. To determine inhaled albuterol and sub-lingual NTG-induced vasodilation (ΔQaw) before, and 30 min and 120 min after a single medium dose of an ICS (220 μg fluticasone) in stable glucocorticoid- naïve COPD patients.

For both aims, the protocol design will be placebo-controlled and double-blind. For the second aim, only fluticasone pretreatment will be possible because the salmeterol component of the fluticasone/salmeterol combination preparation could influence albuterol responsiveness irrespective of any glucocorticoid effect. The timing of the endothelial function measurements in the long-term glucocorticoid/long-acting beta-agonist protocol and single dose ICS protocol is based on the past experience with ICS on airway vascular function. Single dose effects were seen within 15-30 min and waned by 90 min (25,26), while long-term treatment effects were no longer seen 3 weeks after ICS withdrawal (16).

ELIGIBILITY:
Inclusion Criteria:

* Smoking history of at least 10 pack-years and to have quit smoking at least 1 year before the study. -Diagnosis of COPD
* Post-bronchodilator FEV1 of less than 75% of predicted and FEV1/FVC ratio less than 0.7 (GOLD stage ≥2).
* At entry into the study, the subjects will have to be clinically stable; they will be allowed to use short-acting and long-acting β2 - adrenergic agonists and cholinergic antagonists as their usual airway medication.

Exclusion Criteria:

* Women of childbearing potential who do not use accepted birth control measures; pregnant and breast feeding women.
* Use of cardiovascular medications that cannot be held on the study days
* Use of oral airway medications or anti-inflammatory agents
* Subjects with known beta-adrenergic agonist or NTG intolerance
* Acute respiratory infection within four weeks prior to the study
* A body mass index > 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
long term effect of a glucocorticoid/long-acting beta-agonist on endothelial function in the bronchial artery. | 3 weeks
  To determine the effect of a medium dose glucocorticoid/long-acting beta-agonist preparation (250 μg fluticasone plus 50 μg salmeterol) or placebo administered for 3 weeks on inhaled albuterol and sub-lingual NTG induced vasodilation in the bronchial artery, as assessed by ΔQaw in stable glucocorticoid-naïve COPD patients, and to re-assess the responses after a 3 week washout period.

SECONDARY OUTCOMES:
acute effect of an ICS on bronchial endothelial function in stable glucocorticoid-naïve COPD patient. | 30 minutes and 120 minutes after inhaled albuterol and sub-lingual NTG
  To determine inhaled albuterol and sub-lingual NTG-induced vasodilation (ΔQaw) before, and 30 min and 120 minutes after a single medium dose of an ICS (220 μg fluticasone)or placebo in stable glucocorticoid-naïve COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States